CLINICAL TRIAL: NCT06065943
Title: Department of Cardiology Wuerzburg University
Brief Title: Ultrasound-guided In-plane Puncture of the Femoral Artery
Acronym: PARFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 112/19-sc
Record Dates: First submitted 2023-09-05; First posted 2023-10-04 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Vessel Puncture Site Bleeding
Keywords: ultrasound guided puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guidance (Active Comparator)
  Interventions: Procedure: Ultrasound guidance
- Palpation and Fluoroscopy (Other)
  Interventions: Other: Palpation and Fluoroscopy

INTERVENTIONS:
Other: Palpation and Fluoroscopy — Vessel puncture guided palpation and fluoroscopy only
  Arms: Palpation and Fluoroscopy
Procedure: Ultrasound guidance — Vessel puncture guided by Ultrasound
  Arms: Ultrasound guidance

SUMMARY:
In Germany almost 1 million cardiac catheterizations are performed each year. These procedures can be done either by a transradial or a transfemoral approach. Today, the transradial approach is the recommended default strategy. Nevertheless, transfemoral access ist still frequently used. The main draw-back of a transfemoral approach are potential access site complications, which can sometimes be life-threatening. To reduce vascular complications ultrasound guided vessel puncture may be helpful.

In the "Ultrasound guided puncture of the femoral artery"-Study (US-Parfem) an optimized method of ultrasound guided femoral puncture will be evaluated. In this randomized study the new puncture technique combining ultrasound and fluoroscopy will be compared with the conventional method guided by vessel palpation and fluoroscopy. Primary endpoint of the study is the rate of primary successful puncture of the femoral common artery above the bifurcation and below the inguinal ligament ("first success rate").

ELIGIBILITY:
Inclusion Criteria:

* transfemoral catheterization

Exclusion Criteria:

* acute myocardial infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Initial successful puncture of the common femoral artery | 1 week
  Analysis of rotational femoral angiography

SECONDARY OUTCOMES:
Unsuccessful puncture attempts | access-phase of the procedure
  number of unsuccessful puncture attempts
Perception of pain | Evaluated at the end of the access-phase of the procedure
  pain scale between 0 (no pain) and 10 (maximum pain) graded by the patient
accidental venipuncture | at the end of the access-phase of the procedure
  Venipuncture was recognized by backflow of pulsatile and non-arterial blood
Duration until successful puncture | Evaluated at the end of the access-phase of the procedure
  Time frame between start of initial puncture and successful introduction of the guide-wire up to 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voelker W, Lachmann M, Gueder G, Bayik A, Heinrichs M, Kickuth R, Bauer WR, Lengenfelder B, Nordbeck P, Frantz S, Stork S. Can Ultrasound-Guided in-Plane Puncture Technique Enhance the Precision of Femoral Artery Access? The Randomized PARFEM Trial. Catheter Cardiovasc Interv. 2025 Oct;106(4):2252-2262. doi: 10.1002/ccd.31733. Epub 2025 Jul 30. PMID 40735901